CLINICAL TRIAL: NCT00041483
Title: Phase 3 Study to Evaluate Anecortave Acetate vs. Visudyne for the Treatment of the Wet Form of AMD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-01-99
Record Dates: First submitted 2002-07-09; First posted 2002-08-01 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2008-07

CONDITIONS: Macular Degeneration
Keywords: AMD; age-related macular degeneration; Anecortave; Acetate; Wet form of age-related macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — anecortave acetate; Photochemotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Anecortave and Sham PDT (Active Comparator)
  Interventions: Drug: Anecortave Acetate 15 mg sterile suspension; Other: Photodynamic Therapy (PDT)
- PDT and Sham Anecortave Acetate (Active Comparator)
  Interventions: Drug: Anecortave Acetate 15 mg sterile suspension; Other: Photodynamic Therapy (PDT)

INTERVENTIONS:
Drug: Anecortave Acetate 15 mg sterile suspension
Other: Photodynamic Therapy (PDT)

SUMMARY:
The purpose of this study is to demonstrate that Anecortave Acetate is as effective after twelve months of treatment as photodynamic therapy (PDT) with Visudyne in patients eligible for initial PDT treatment for wet age-related macular degeneration.

ELIGIBILITY:
Patients of any race, either gender, aged 50 years and above, diagnosed with subfoveal CNV due to AMD with best corrected logMAR visual acuity of 20/40 (snellen equivalent) to 20/400 (Snellen equivalent) in the study eye. Clinically relevant concomitant diseases will be excluded.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2002-06; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Percentage of Patients Maintaining Vision | Month 12

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States